CLINICAL TRIAL: NCT04742114
Title: Effect of EPAP Device on Emphysema and Lung Bullae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QiluH 2020039123
Record Dates: First submitted 2021-01-21; First posted 2021-02-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Emphysema; Bullous Disease Lung
Keywords: Emphysema; Bullous; Expiratory Positive Airway Pressure
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Intervention Model Description: The subjects were divided into two groups. The first group use the breathing mask without the positive pressure valve, and the second group use the breathing mask with a positive pressure valve, that is EPAP breathing mask.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the face mask without EPAP (Sham Comparator): Will be collected clinical and anthropometric data of the participant. Will have the pulmonary function test every two months. Will be collected CT scan data. Patients will conduct 6MWT every two months. Borg scale data will be collected.The face mask without the application of EPAP will be used.
  Interventions: Device: use the face mask without Expiratory Positive Airway Pressure(EPAP).
- the face mask with EPAP (Experimental): Will be collected clinical and anthropometric data of the participant. Will have the pulmonary function test every two months. Will be collected CT scan data. Patients will conduct 6MWT every two months. Borg scale data will be collected.The application of EPAP (15cmH2O) via face mask will be used.
  Interventions: Device: use the face mask with Expiratory Positive Airway Pressure(EPAP).

INTERVENTIONS:
Device: use the face mask with Expiratory Positive Airway Pressure(EPAP). — The subjects were divided into two groups. The first group use the face mask without EPAP, and the other group use the face mask with EPAP.
  Arms: the face mask with EPAP
Device: use the face mask without Expiratory Positive Airway Pressure(EPAP). — The subjects were divided into two groups. The first group use the face mask without EPAP, and the other group use the face mask with EPAP.
  Arms: the face mask without EPAP

SUMMARY:
The purpose of this study is to evaluate the safety and the effects and of the application of Expiratory Positive Airway Pressure (EPAP) device on Dynamic Hyperinflation and dyspnea in patients with Emphysema and pulmonary bullae.

DETAILED DESCRIPTION:
The trial will last for six months. Patients will be collected clinical and anthropometric data by using questionnaires initially. Patients will have the pulmonary function test and CT scan and conduct 6MWT every two months. And Borg scale data will be collected every two months. The application of EPAP (15cmH2O) via face mask will be randomized with the help of opaque envelopes.

ELIGIBILITY:
Inclusion Criteria:

* The patient was ≤75 years old
* CT examination revealed emphysema (absolute CT value ≥900) or bullae
* CT do not show other imaging changes of lung diseases, such as mass, exudation and interstitial changes
* No history of lung cancer, pneumonectomy, any history of cystic fibrosis, allergic alveolitis, or pulmonary fibrosis
* Patients volunteer to participate and sign informed consent

Exclusion Criteria:

* Patients with asthma, bronchiectasis, interstitial lung disease and other basic lung diseases
* Patients with heart failure
* Patients with a history of malignancy
* Patients are reluctant to participate

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
CT DICOM data | Change from Baseline CT attenuation value at 6 months.
  Quantitative analysis of emphysema severity will be performed on segmented lung images by using the Slicer software package. The total emphysema percentage will be defined as all lung voxels with a CT attenuation value of less than - 910 HU.

SECONDARY OUTCOMES:
FVC in pulmonary function test | Change from Baseline FVC data at 2 months.
  The data of the patient's FVC will be collected to evaluate the change of the patient's lung function.
FVC in pulmonary function test | Change from Baseline FVC data at 4 months.
  The data of the patient's FVC will be collected to evaluate the change of the patient's lung function.
FVC in pulmonary function test | Change from Baseline FVC data at 6 months.
  The data of the patient's FVC will be collected to evaluate the change of the patient's lung function.
FVC% in pulmonary function test | Change from Baseline FVC% data at 2 months.
  The data of the patient's FVC% will be collected to evaluate the change of the patient's lung function.
FVC% in pulmonary function test | Change from Baseline FVC% data at 4 months.
  The data of the patient's FVC% will be collected to evaluate the change of the patient's lung function.
FVC% in pulmonary function test | Change from Baseline FVC% data at 6 months.
  The data of the patient's FVC% will be collected to evaluate the change of the patient's lung function.
FEV1 in pulmonary function test | Change from Baseline FEV1 data at 2 months.
  The data of the patient's FEV1 will be collected to evaluate the change of the patient's lung function.
FEV1 in pulmonary function test | Change from Baseline FEV1 data at 4 months.
  The data of the patient's FEV1 will be collected to evaluate the change of the patient's lung function.
FEV1 in pulmonary function test | Change from Baseline FEV1 data at 6 months.
  The data of the patient's FEV1 will be collected to evaluate the change of the patient's lung function.
FEV1% in pulmonary function test | Change from Baseline FEV1% data at 2 months.
  The data of the patient's FEV1% will be collected to evaluate the change of the patient's lung function.
FEV1% in pulmonary function test | Change from Baseline FEV1% data at 4 months.
  The data of the patient's FEV1% will be collected to evaluate the change of the patient's lung function.
FEV1% in pulmonary function test | Change from Baseline FEV1% data at 6 months.
  The data of the patient's FEV1% will be collected to evaluate the change of the patient's lung function.
FEV1/ FVC% in pulmonary function test | Change from Baseline FEV1/ FVC% data at 2 months.
  The data of the patient's FEV1/ FVC% will be collected to evaluate the change of the patient's lung function.
FEV1/ FVC% in pulmonary function test | Change from Baseline FEV1/ FVC% data at 4 months.
  The data of the patient's FEV1/ FVC% will be collected to evaluate the change of the patient's lung function.
FEV1/ FVC% in pulmonary function test | Change from Baseline FEV1/ FVC% data at 6 months.
  The data of the patient's FEV1/ FVC% will be collected to evaluate the change of the patient's lung function.
TLC in pulmonary function test | Change from Baseline TLC data at 2 months.
  The data of the patient's TLC will be collected to evaluate the change of the patient's lung function.
TLC in pulmonary function test | Change from Baseline TLC data at 4 months.
  The data of the patient's TLC will be collected to evaluate the change of the patient's lung function.
TLC in pulmonary function test | Change from Baseline TLC data at 6 months.
  The data of the patient's TLC will be collected to evaluate the change of the patient's lung function.
RV/TLC in pulmonary function test | Change from Baseline RV/TLC data at 2 months.
  The data of the patient's RV/TLC will be collected to evaluate the change of the patient's lung function.
RV/TLC in pulmonary function test | Change from Baseline RV/TLC data at 4 months.
  The data of the patient's RV/TLC will be collected to evaluate the change of the patient's lung function.
RV/TLC in pulmonary function test | Change from Baseline RV/TLC data at 6 months.
  The data of the patient's RV/TLC will be collected to evaluate the change of the patient's lung function.
FRC in pulmonary function test | Change from Baseline FRC data at 2 months.
  The data of the patient's FRC will be collected to evaluate the change of the patient's lung function.
FRC in pulmonary function test | Change from Baseline FRC data at 4 months.
  The data of the patient's FRC will be collected to evaluate the change of the patient's lung function.
FRC in pulmonary function test | Change from Baseline FRC data at 6 months.
  The data of the patient's FRC will be collected to evaluate the change of the patient's lung function.
ETCO2 | Change from Baseline ETCO2 data at 2 months during the intervention.
  ETCO2 data will be collected to assess changes in CO2 retention in patients.
ETCO2 | Change from Baseline ETCO2 data at 4 months during the intervention.
  ETCO2 data will be collected to assess changes in CO2 retention in patients.
ETCO2 | Change from Baseline ETCO2 data at 6 months during the intervention.
  ETCO2 data will be collected to assess changes in CO2 retention in patients.
6 minutes walk test(6MWT) | Change from Baseline 6MWT data at 2 months during the intervention.
  The 6 minutes walk test data will be collected to assess the cardiopulmonary function of the patients
6 minutes walk test(6MWT) | Change from Baseline 6MWT data at 4 months during the intervention.
  The 6 minutes walk test data will be collected to assess the cardiopulmonary function of the patients
6 minutes walk test(6MWT) | Change from Baseline 6MWT data at 6 months during the intervention.
  The 6 minutes walk test data will be collected to assess the cardiopulmonary function of the patients
Borg scale score | Change from Baseline Borg scale score data at 2 months during the intervention.
  The Borg scale data will be collected to assess changes in dyspnea.The scale scores range from 0 to 10, with 0 indicating the minimum and 10 indicating the maximum. The higher the score, the more severe the dyspnea is.
Borg scale score | Change from Baseline Borg scale score data at 4 months during the intervention.
  The Borg scale data will be collected to assess changes in dyspnea.The scale scores range from 0 to 10, with 0 indicating the minimum and 10 indicating the maximum. The higher the score, the more severe the dyspnea is.
Borg scale score | Change from Baseline Borg scale score data at 6 months during the intervention.
  The Borg scale data will be collected to assess changes in dyspnea.The scale scores range from 0 to 10, with 0 indicating the minimum and 10 indicating the maximum. The higher the score, the more severe the dyspnea is.

CONTACTS AND LOCATIONS:
Overall Officials: dedong ma, Doctor, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Background] Ranieri VM, Giuliani R, Cinnella G, Pesce C, Brienza N, Ippolito EL, Pomo V, Fiore T, Gottfried SB, Brienza A. Physiologic effects of positive end-expiratory pressure in patients with chronic obstructive pulmonary disease during acute ventilatory failure and controlled mechanical ventilation. Am Rev Respir Dis. 1993 Jan;147(1):5-13. doi: 10.1164/ajrccm/147.1.5. PMID 8420430
- [Background] Fagevik Olsen M, Lannefors L, Westerdahl E. Positive expiratory pressure - Common clinical applications and physiological effects. Respir Med. 2015 Mar;109(3):297-307. doi: 10.1016/j.rmed.2014.11.003. Epub 2014 Nov 12. PMID 25573419
- [Background] Blanch L, Bernabe F, Lucangelo U. Measurement of air trapping, intrinsic positive end-expiratory pressure, and dynamic hyperinflation in mechanically ventilated patients. Respir Care. 2005 Jan;50(1):110-23; discussion 123-4. PMID 15636649
- [Background] Kondili E, Alexopoulou C, Prinianakis G, Xirouchaki N, Georgopoulos D. Pattern of lung emptying and expiratory resistance in mechanically ventilated patients with chronic obstructive pulmonary disease. Intensive Care Med. 2004 Jul;30(7):1311-8. doi: 10.1007/s00134-004-2255-z. Epub 2004 Mar 31. PMID 15054570
- [Background] Gosselink R. Controlled breathing and dyspnea in patients with chronic obstructive pulmonary disease (COPD). J Rehabil Res Dev. 2003 Sep-Oct;40(5 Suppl 2):25-33. doi: 10.1682/jrrd.2003.10.0025. PMID 15074451
- [Background] Dechman G, Wilson CR. Evidence underlying breathing retraining in people with stable chronic obstructive pulmonary disease. Phys Ther. 2004 Dec;84(12):1189-97. PMID 15563259
- [Background] Puente-Maestu L, Stringer WW. Hyperinflation and its management in COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(4):381-400. doi: 10.2147/copd.2006.1.4.381. PMID 18044095
- [Derived] Xu Z, Han Z, Ma D. Efficacy and safety of long-term use of a positive expiratory pressure device in chronic obstructive pulmonary disease patients, a randomized controlled trial. BMC Pulm Med. 2023 Jan 16;23(1):17. doi: 10.1186/s12890-023-02319-5. PMID 36647057